CLINICAL TRIAL: NCT00236600
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Efficacy and Safety of Topiramate in Weight Loss Maintenance in Obese Patients Following Participation in an Intensive, Non-Pharmacologic Weight Loss Program
Brief Title: A Study on Efficacy and Safety of Topiramate in Maintaining Weight Loss in Obese Patients Following an Intensive, Non-Pharmacologic Weight Loss Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003706
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Obesity; Hypertension; Hyperlipidemia; Type 2 Diabetes; Life style modification
MeSH Terms: conditions — Obesity; Hypertension; Hyperlipidemias; Diabetes Mellitus, Type 2 | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of topiramate 96mg and 192mg daily) with placebo in the treatment of obesity following an intensive non-pharmacologic weight loss program.

DETAILED DESCRIPTION:
Although dietary modification coupled with increased exercise is the preferred treatment of obesity, these lifestyle changes alone are often insufficient in achieving and maintaining weight reduction in obese patients. Topiramate is not approved for the treatment of obesity. This double-blind, placebo controlled study will evaluate the effectiveness and safety of topiramate in maintaining weight loss achieved by an intensive non-drug weight reduction program. Enrolled patients will undergo run-in phase (8 weeks of intensive non-drug weight reduction therapy consisting of a low calorie diet, a behavioral modification program, and an exercise program). Those patients who achieve weight loss of >= 8% of enrollment body weight and meeting the eligibility criteria will be randomized to either 96mg or 192mg of topiramate, or placebo. After 8 weeks of dose titration, the patients will receive one year of treatment. Effectiveness will be assessed by body weight, Body Mass Index (BMI), number and proportion of 5%, 10% and 15% weight loss responders, number and proportion of patients who maintain 50%, 75%, and 100% of weight lost during run-in phase, waist and hip circumferences, fasting lipid profile, fasting plasma glucose, HbA1c, fasting insulin, two-hour glucose tolerance test, uric acid level, blood pressure, body composition, echocardiography, and Health Related Quality of Life scores. Safety evaluations (incidence of adverse events, electrocardiograms, vital signs, etc) will be performed throughout the study. The study hypothesis is that topiramate is more effective than placebo in maintaining weight reduction in obese patients following intensive non-drug weight reduction program. During the initial 8 weeks, the doses of topiramate or placebo will be gradually increased to the target doses (either 96mg or 192mg) daily by mouth and the doses will be maintained for one year.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >= 33 and < 50 kg/m2
* BMI >=30 and < 50 kg/m2 if patients have controlled hypertension or abnormal blood lipids
* Stable weight
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing abstinence, or practicing an acceptable method of contraception (requires negative pregnancy test)
* Randomization criteria: Weight reduction of more than 8% of enrollment body weight during the eight week run-in phase

Exclusion Criteria:

* Prior exposure, known contraindication, or hypersensitivity to topiramate
* Exposure to any other experimental drug or device within last 30 days
* A diagnosis of diabetes (except those diagnosed during the enrollment if no medications are needed)
* History or evidence of clinically significant liver disease, cardiovascular disease, uncontrolled hypertension or high thyroid levels
* History of obesity with known cause
* History or family history of kidney stones
* History of weight loss surgery or liposuction
* History of malignancy within last 5 years
* History of an eating disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2000-08; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight from the enrollment visit to week 60.

SECONDARY OUTCOMES:
Change from baseline to week 60 in absolute change in body weight, body mass index, waist circumference, fasting lipid profile; safety evaluations over study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Astrup A, Caterson I, Zelissen P, Guy-Grand B, Carruba M, Levy B, Sun X, Fitchet M. Topiramate: long-term maintenance of weight loss induced by a low-calorie diet in obese subjects. Obes Res. 2004 Oct;12(10):1658-69. doi: 10.1038/oby.2004.206. PMID 15536230